CLINICAL TRIAL: NCT02027181
Title: Automation of the Oxygen's Administration in Spontaneous Ventilation (FreeO2) During the Hypoxemic Acute Respiratory Distress
Brief Title: Automatic Administration of Oxygen During Respiratory Distress
Acronym: FreeO2-Hypox
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RB 10-071 FreeO2-Hypox
Record Dates: First submitted 2013-10-17; First posted 2014-01-06 (Estimated); Last update posted 2014-10-31 (Estimated); Status verified 2014-10

CONDITIONS: Acute Respiratory Distress Syndrome; Hypoxemia
MeSH Terms: conditions — Respiratory Distress Syndrome; Hypoxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- device FreeO2 (Experimental): Automatic adjustment of oxygen
  Interventions: Device: Device FreeO2 v2.0
- Manual oxygenation (Active Comparator): Manual adjustment of oxygen
  Interventions: Device: Device FreeO2 v2.0

INTERVENTIONS:
Device: Device FreeO2 v2.0 — * Automatic adjustment of oxygen through the "Free O2" device.
  * "FreeO2" device in mode medical data collecting(SpO2,EtCO2...).
  Arms: device FreeO2
Device: Device FreeO2 v2.0 — * Manual adjustment of oxygen without the assistance of the "FreeO2" device.
  * Only "FreeO2" device in mode medical data collecting(SpO2,EtCO2...).
  Arms: Manual oxygenation

SUMMARY:
Aim: The purpose of this study is to evaluate the use feasibility of FreeO2 so as to deliver automatically oxygen in the emergency department in a patient population admitted for acute respiratory failure.

Hypothesis: The principal hypothesis is that FreeO2 is possible and well-accepted by nurses and medical personnel and there are advantages to use this system. In comparison with the common oxygen delivery (the rotameter), the hypothesis is that FreeO2 system will make for a better control of the oxygen saturation in function of designed target, reducing the desaturation time and hyperoxia. We think that oxygen weaning will be faster than classical way if it is automated. In addition, FreeO2 could reduce the number of intervention by nurse personnel.

ELIGIBILITY:
Inclusion Criteria:

* Admission to the emergency for respiratory disease (or cardiac - acute pulmonary edema)justifying an oxygen administration to over 3 L / min to maintain a SpO2 ≥ 92%.
* Inclusion within a time less than two hours after the start of the oxygen at the emergency.
* Patient consent,or a close.

Exclusion Criteria:

* Necessity of an oxygen flow exceeds 15 L / min to maintain a SpO2 higher than 92%.
* Criteria of gravity justifying immediately a different technique of ventilatory support:
* Disturbance of consciousness with a Glasgow Coma Score ≤ 12
* Serious ventricular rhythm disorders
* Hemodynamic instability (SBP <80mmHg or recourse to vasopressors)
* Cardiac or respiratory arrest
* pH < 7.35 and PaCO2 > 55 mm Hg
* Necessity of a urgent surgery, or coronary revascularization
* Age <18 years
* Pregnant women, lactating
* Patient not relevant
* Unavailability of the prototype FreeO2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2011-08; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Percentage of time spent in the target zone of oxygen saturation in the acute phase of treatment | 3 hours or 1 hour after after cessation of oxygenation
  The target zone of oxygen saturation is : SpO2 = 92-96% The "acute phase of treatment" is defined by the 3 first hours of treatment by oxygenation and/or until one hour after the end of this last.

SECONDARY OUTCOMES:
nursing workload assessed by the number of manual Oxygen flow adjustments and airway management procedures | 3 days max
Time spent in a area of severe desaturation (SpO2 <88%) and a hyperoxia area (SpO2> 98%). | 3 hours or 1 hour after after cessation of oxygenation
Maintaining EtCO2 in a selected area | 3 hours or 1 hour after after cessation of oxygenation
Oxygen consumption measured at the end of administration | 3 hours or 1 hour after after cessation of oxygenation
Duration of administration during hospitalization | 28 days max
Number of complications related to the administration of oxygen | 28 days max
Frequency of use of invasive or noninvasive ventilation during hospitalization. | 28 days max

CONTACTS AND LOCATIONS:
Overall Officials: Erwan L'HER, Principal Investigator — University Hospital, Brest
Locations (4):
- Canada (2):
  - Hopital Hotel Dieux de Levis, Lévis, Quebec
  - Institut universitaire de Cardiologie et de Pneumologie de Québec, Québec, Quebec
- France (2):
  - HIA Clermont Tonnerre, Brest
  - Brest, University Hospital, Brest

REFERENCES:
- [Derived] L'Her E, Dias P, Gouillou M, Riou A, Souquiere L, Paleiron N, Archambault P, Bouchard PA, Lellouche F. Automatic versus manual oxygen administration in the emergency department. Eur Respir J. 2017 Jul 20;50(1):1602552. doi: 10.1183/13993003.02552-2016. Print 2017 Jul. PMID 28729473